CLINICAL TRIAL: NCT07263698
Title: Investigation of Clinical Efficacy of a New Mouthwash on Reducing Dental Plaque and Helping Prevent Gum Problems as Compared to a Control Mouthwash - a Three-month Study in Italy
Brief Title: Investigation of Clinical Efficacy of a New Mouthwash on Reducing Dental Plaque and Helping Prevent Gum Problems as Compared to a Control Mouthwash
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2025-10-PGN-PRG-ITA-YPZ
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Gingivitis; Plaque, Dental
Keywords: Quigley-Hein Plaque Index; Modified Gingival
MeSH Terms: conditions — Gingivitis; Dental Plaque | interventions — Cetylpyridinium; cytidylyl-(3'-5')-cytidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test 1 mouthwash (Experimental): After brushing in the morning and in the evening, 20 ml of mouthwash shall be used for each rinsing, 2 times daily (morning and evening) for 30 seconds each time. No further rinsing with water shall be occurred after each mouthwash rising. Each qualified subject will follow this specific application for 3 months
  Interventions: Drug: cetylpyridinium chloride (CPC), zinc lactate and sodium fluoride Mouthwash
- Test 2 mouthwash (Active Comparator): After brushing either in the morning or in the evening, 20 ml of the mouthwash shall be used for each rinsing, 2 times daily (morning and evening) for 30 seconds each time
  Interventions: Drug: sodium fluoride Mouthwash

INTERVENTIONS:
Drug: cetylpyridinium chloride (CPC), zinc lactate and sodium fluoride Mouthwash — 0.09% CPC, 0.28% zinc lactate and 500 ppm F as sodium fluoride
  Arms: Test 1 mouthwash
Drug: sodium fluoride Mouthwash — 100 ppm F as sodium fluoride
  Arms: Test 2 mouthwash

SUMMARY:
Qualified subjects will be enrolled and randomized to either one of the two study groups described above based on their initial modified gingivitis and plaque scores. Subjects will be instructed to use the products according to the instructions provided. Subjects will return to the dental office for evaluation after two weeks, six weeks and three months of product use. All subjects will be followed for adverse events throughout the study

ELIGIBILITY:
Inclusion Criteria:

* Subjects, ages 18-70, inclusive.
* Availability for the three-month duration of the clinical research study.
* Good general health.
* Initial modified gingivitis index of at least 1.5 as determined by the use of the Modified Gingival Index.
* Initial plaque index of at least 1.5 as determined by the use of the Quigley-Hein Plaque Index.
* Signed Informed Consent Form (Appendix C)

Exclusion Criteria:

* Presence of orthodontic bands.
* Tumor(s) of the soft or hard tissues of the oral cavity.
* Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone).
* Five or more carious lesions requiring immediate restorative treatment.
* Antibiotic use any time during the one-month period prior to entry into the study.
* Participation in any other clinical study or test panel within the one month prior to entry into the study.
* Dental prophylaxis during the past two weeks prior to baseline examinations.
* History of allergies to oral care/personal care consumer products or their ingredients.
* On any prescription medicines that might interfere with the study outcome.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Modified Gingival Index | baseline, 2 week, 6 week & 3 month
  A Modified Gingivitis Index score from 0 to 4 will be assigned by the examiner to all tooth surfaces. In regards to the scale, lower number is a better outcome.
Saxton Bleeding Index | baseline, 2 week, 6 week & 3 month
  Gingival bleeding is assessed 30 seconds after probing; a score of 0 represents an absence of bleeding.
  a score of 1 is given if bleeding is observed within 30 seconds after probing and a score of 2 is given if bleeding is observed immediately on probing
Modified Quigley-Hein Plaque Index | baseline, 2 week, 6 week & 3 month
  Modified Quigley-Hein Plaque Index score of 0 to 5 will be assigned to all scoreable disclosed tooth surfaces. In regards to the scale, lower number is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Montesani, DDS, Principal Investigator — University of Rome
Locations (1):
- Clinica Odontoiatrica Montesani, Roma, Rome, Italy